CLINICAL TRIAL: NCT03252054
Title: Prevalence of Memory and Attention Disorders and Malnutrition in Hospitalized Older Adults (Muistitoimintojen ja Tarkkaavaisuuden häiriöiden ja Vajaaravitsemuksen Yleisyys iäkkäillä Sairaalahoidossa Olevilla Potilailla [Finnish])
Brief Title: Memory and Attention Disorders and Malnutrition in Hospital Setting
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Coxa, Hospital for Joint Replacement (Other); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: Ger1-16
Record Dates: First submitted 2017-08-09; First posted 2017-08-17 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Dementia; Delirium; Cognitive Impairment; Malnutrition
MeSH Terms: conditions — Dementia; Delirium; Cognitive Dysfunction; Malnutrition | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 70 or over: Patients eligible for the study will undergo screening for memory disorders, attention disorders, and malnutrition
  Interventions: Diagnostic Test: Screening for memory disorders, attention disorders, and malnutrition

INTERVENTIONS:
Diagnostic Test: Screening for memory disorders, attention disorders, and malnutrition — Screening for memory disorders, attention disorders, and malnutrition, using Six-Item Screener, Months of the Year Backwards Test, and NRS-2002 and MNA-SF, respectively.

SUMMARY:
This is a cross-sectional observational study that investigates the prevalence of memory disorders, attention disorders (suggesting delirium), and malnutrition in hospitalized older adults (aged 70 years or over) in a tertiary care centre, using rapid screening toos (Six-item screener for memory disorders, Months of the Year Backwards Test for delirium, and NRS-2002 and Mini Nutritional Assessment Short Form for malnutrition).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in Tampere University Hospital (excl. psyciatry, pediatrics, ICU)
* Able to communicate in Finnish

Exclusion Criteria:

* Unable to communicate because of unconciuousness, critical health status, or communication difficulties
* Having a (surgical) procedure at the time of data collection

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients born in 1946 or earlier hospitalized in somatic wards.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of memory disorders | day of recruitment
  Abnormal result in Six-Item Screener
Prevalence of attention disorders | day of recruitment
  Abnormal result in Months of the Year Backwards Test
Prevalence of malnutrition and risk of malnutrition | day of recruitment
  Abnormal result based on nutritional status screening tools

CONTACTS AND LOCATIONS:
Overall Officials: Esa Jämsen, MD, PhD, Study Director — consultant

IPD SHARING:
Plan to Share IPD: No